CLINICAL TRIAL: NCT02199756
Title: Development of Nanovectors to Prevent Placental Passage of a Tocolytic Agent
Brief Title: Nanovectors to Prevent Placental Passage of Tocolytic Agents
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Jerrie Refuerzo, Associate Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-14-0370
Record Dates: First submitted 2014-07-23; First posted 2014-07-24 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-11

CONDITIONS: Preterm Labor
Keywords: Uterine contractions; Indomethacin; Nanovectors
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Uterine biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cesarean section: Women with cesarean section

SUMMARY:
The purpose of the study is to find out whether indomethacin encapsulated within a nanovector can stop contractions in pregnant human uterine tissue. Preterm delivery is a major contributor to newborn deaths. The treatment of preterm labor includes medications that stop contractions within the uterus, or womb. Indomethacin is effective in stopping uterine contractions, but crosses the placenta to the unborn baby causing problems for the baby. Nanovectors are used to direct the delivery of medications. If indomethacin can be delivered directly to the uterus using a nanovector, it may be an ideal medication to treat preterm labor. We hypothesize that nanovectors loaded with indomethacin will reduce uterine contractions.

DETAILED DESCRIPTION:
This is a prospective observational study.

Subjects will undergo a biopsy from the middle of the upper margin of the uterine incision measuring 4 x 2 x 2 cm. This will be performed by the managing doctor at the time of cesarean section after delivery of the baby. Once the tissue is obtained, the site will be closed using sutures similar to the usual closure of the uterus at cesarean section. This biopsy will be taken to the laboratory to test whether the nanovector will increase or decrease contractions in the uterus. Once this test is finished, the tissue will be frozen and test for the absence or presence of the nanovector within the tissue.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women undergoing elective cesarean section who are greater than 37 weeks

Exclusion Criteria:

* Known infection

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women who will undergo elective cesarean section at term
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2014-07; Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Uterine contractions | 3 hours
  Uterine biopsies obtained from subjects will be placed in a specimen chamber that measures uterine contractility. Mean contractile intensity will be determined before and after exposure to oxytocin, indomethacin, liposomes and liposome indomethacin.

CONTACTS AND LOCATIONS:
Overall Officials: Jerrie S Refuerzo, M.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Hospital Texas Medical Center, Houston, Texas, United States